CLINICAL TRIAL: NCT00203385
Title: Maintenance Phase Treatment With Divalproex for Post Traumatic Stress Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding expired
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Responsible Party: Principal Investigator, Lori Davis, MD, Associate Chief of Staff, Tuscaloosa Research & Education Advancement Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREAC Maintenance DVX PTSD
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: PTSD
Keywords: divalproex sodium, depakote, ptsd, long-term ptsd treatments
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Valproic Acid

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Divalproex (Experimental): Divalproex; oral up to 2000mg/d; open label
  Interventions: Drug: Divalproex

INTERVENTIONS:
Drug: Divalproex — Depakote up to 2000mg/d
  Other Names: Depakote

SUMMARY:
The primary objective is to evaluate the long-term efficacy of divalproex sodium (Depakote) in the continuation treatment of PTSD.

DETAILED DESCRIPTION:
Patients who have participated in the 8-week randomized, double-blind, placebo-controlled treatment trial of divalproex for PTSD and have signed informed consent will be enrolled in a 24-week open-label divalproex continuation phase trial. Patients' symptoms, side effects and compliance will be assessed every two weeks for 4 weeks, then every 4 weeks, thereafter, up to 24-weeks. Based on symptomology and occurrence of side effects, the investigator will titrate the medication in 500 mg (one tablet) increments every four days, as tolerated, until a maximum therapeutic benefit is achieved, not to exceed 3000 mg/day. The dosing is twice daily, with the higher dose at bedtime. Compliance will be assessed by monthly pill count and valproic acid levels at the week(s) 4, 12 and 24. Patients are given supportive clinical management during the clinic visits. An investigator is available by telephone 24 hrs a day in case of emergency. Patients may be seen more often if needed. Efficacy will be measured by the structured rating scales for depression, global function and assessment and PTSD. Results of this study will be used to evaluate the long-term efficacy of divalproex in the maintenance treatment of PTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PTSD, confirmed by MINI and CAPS.
2. Participation in the placebo-controlled acute phase study with divalproex for PTSD
3. Age 19 or older
4. No substance abuse/dependence for the previous 6 weeks (except for nicotine and caffeine)
5. Clinically normal physical and laboratory examination (lab profile listed below). LFTs up to 2.5 times the normal limit will be allowed.
6. Women of childbearing potential must be using medically approved methods of birth control (such as a condom, birth control pill, DepoProvera, or diaphragm with spermicide)
7. Signed informed consent
8. Male or female, any race or ethic origin

Exclusion Criteria:

1. Lifetime history of bipolar I, psychotic, or cognitive disorders
2. Actively suicidal, homicidal, or psychotic
3. History of sensitivity to divalproex
4. Unstable general medical conditions
5. Score ≥ 6 on Question #10 of MADRS
6. Women who are pregnant, planning to become pregnant or breastfeed during the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-05 (Actual); Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | 24 weeks
  Clinician-administered rating scale to assess PTSD, 17-items, higher score is more severe, range from zero to 136

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale Subscores | 24 weeks
  Clinician-administered rating scale to assess PTSD clusters of re-experiencing, avoidance and emotional numbing, and hyperarousal; higher score is more severe.

CONTACTS AND LOCATIONS:
Overall Officials: Lori L Davis, MD, Principal Investigator — Tuscaloosa Veterans Affairs Medical Center
Locations (1):
- Tuscaloosa Research & Education Advancement Corporation, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark RD, Canive JM, Calais LA, Qualls CR, Tuason VB. Divalproex in posttraumatic stress disorder: an open-label clinical trial. J Trauma Stress. 1999 Apr;12(2):395-401. doi: 10.1023/A:1024797014210. PMID 10378177